CLINICAL TRIAL: NCT03660787
Title: Phase II Multi-center Randomized Double-blind Placebo-controlled Efficacy and Dose Ranging Trial of the Drug Product Seroguard, Solution (JSC Pharmasyntez, Russia) Used for the Prevention of Pelvic Adhesions
Brief Title: Efficacy and Dose Ranging Study of Seroguard
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmasyntez (Industry)
Collaborators: Cromos Pharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SG-2/1215
Record Dates: First submitted 2018-08-31; First posted 2018-09-07 (Actual); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Adhesion
Keywords: Adhesion; Efficacy
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The present study was conducted as a double blind trial. Neither a medical investigator, nor patients had access to the treatment assignment code in order to ensure the maximum objective evaluation of the primary endpoint.
  Blinding was performed in such a way that disclosing a randomization code of a certain subject excluded a disclosure of the code in general (i.e. the randomization code had no indication to the treatment group). However, there were no cases of the randomization code disclosure in the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo, 1.5 mL/kg (Placebo Comparator): each subject received the placebo at the dose of 1.5 mL/kg of body weight;
  Interventions: Drug: Placebo
- Placebo, 2.4 mL/kg (Placebo Comparator): each subject received the placebo at the dose of 2.4 mL/kg of body weight;
  Interventions: Drug: Placebo
- Seroguard, 1.5 mL/kg (Experimental): each subject received the test drug at the dose of 1.5 mL/kg of body weight;
  Interventions: Drug: Seroguard
- Seroguard, 2.4 mL/kg (Experimental): each subject received the test drug at the dose of 2.4 mL/kg of body weight.
  Interventions: Drug: Seroguard

INTERVENTIONS:
Drug: Seroguard — Seroguard 0.41 g/L solution
  Arms: Seroguard, 1.5 mL/kg; Seroguard, 2.4 mL/kg
Drug: Placebo — Saline
  Arms: Placebo, 1.5 mL/kg; Placebo, 2.4 mL/kg

SUMMARY:
This trial was a multi-center, double-blind, randomized, parallel group, placebo-controlled, phase II study in adult hospitalized female patients with the confirmed diagnosis of pelvic adhesive disease in Study centres in Russia.

DETAILED DESCRIPTION:
In order to evaluate efficacy and safety of Seroguard, solution for IP administration, a study design meeting the set objectives was selected: prospective, multi-center, double-blind, randomized, parallel group, placebo-controlled study.

Given the fact that comparison with placebo is considered the best way to prove efficacy and safety of a drug and that currently there are no drugs with a similar mechanism of action at the pharmaceutical product market, a placebo-controlled, parallel group study design was selected.

A randomized, parallel group study design was chosen in order to ensure minimization of a selection bias.

Subjects were randomized into four groups (two groups of the test drug and two placebo groups corresponding to the two doses) to enable a comparison of Seroguard administration at two doses.

A double-blind study design was selected in order to ensure minimization of an outcome evaluation bias.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged from 18 to 45 years with the confirmed diagnosis of pelvic adhesions having indications for surgery (laparoscopic adhesiolysis).
2. Voluntarily and personally signed and dated Form of Informed Consent.
3. Female patients with pelvic adhesions confirmed by gynecological and ultrasound examination.

Exclusion Criteria:

1. Female patients having contraindications to surgical treatment (including acute or exacerbated chronical adnexal inflammation);
2. Body mass index of 30.0 kg/m2 and more;
3. Known hypersensitivity to the test drug components (Seroguard);
4. Pregnancy, breastfeeding or planning a pregnancy during the clinical trial;
5. Refusal to use effective contraception methods throughout the study;
6. Positive HIV, RW, HBV or HCV test result;
7. Alcohol abuse, drug addiction, and toxicomania (except smoking);
8. American Society of Anesthesiologists physical status category III and more (ASA);
9. Purulent process in the abdominal cavity;
10. Disseminated endometriosis;
11. WBC count more than 10*109/L at the complete blood count;
12. Need of using any drugs during the surgery other than 0.02% chlorhexidine aqueous solution throughout the surgery, as well as the test drug or the placebo (0.9% sodium chloride) administered intraperitoneally in the end of surgery.
13. Concomitant diseases that may require conversion of the surgical intervention by other indications;
14. Type I or II diabetes mellitus;
15. Deep vein thrombosis and/or PATE at the screening or in the medical history;
16. Renal impairment (glomerular filtration rate less than 60 mL/min/1.73 m2 assessed by the CKD-EPI equation);
17. Liver disorders defined as more than 2-fold rise of the upper limit of normal of one of the following enzymes: ALT, AST, GGTP, AP, or more than 2-fold total bilirubin increase;
18. Myocardial infarction within 6 months before screening;
19. Any concomitant diseases accompanied by heart failure;
20. Clinically significant ECG changes (as to the investigator's opinion);
21. Any concomitant diseases accompanied by respiratory failure;
22. Any oncological disease within 3 years before enrollment into the study;
23. Systemic inflammatory diseases;
24. Diseases associated with chronic hemorrhages;
25. Blood diseases (anemias of any origin, hemoglobinopathies, inherited and acquired coagulopathies, hemostasis disorders, thrombocytopenias, and thrombocytopathias, any hemoblastoses);
26. Any other disease that, in the investigator's opinion, may affect study results or present an additional threat to well-being of a patient after administration of the study drug;
27. Use of anticoagulants, antiaggregants (except for acetylsalicylic acid at the dose of less than 325 mg/day) at the moment of inclusion into the study or planning to do so during the study;
28. Use of drugs with pronounced hemato-, hepato-, or nephrotoxic action, drugs of biological origin;
29. Need to administer cytostatics, systemic glucocorticosteroids, and other immunosuppressive agents during the patient's participation in the study.
30. Participation in any other clinical trial within 30 days before screening;
31. Contraindications to MRI (presence of implants or implanted electronic devices);
32. Impossibility or inability to comply with the requirements of the protocol, including for physical, psychic or social reasons, in the investigator's opinion.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Shurygin, PhD,D.M.Sc., Study Chair — Pharmasyntez
Locations (14):
- Russia (14):
  - Krai Government-Owned State Funded Healthcare Institution "Krai Clinical Hospital", Krasnoyarsk, Krasnoyarsk Krai
  - State Educational Government-Financed Institution of Higher Professional Education "Krasnoyarsk State Medical University named after Prof. V.F. Voino-Yasenetsky" of the Ministry of Healthcare of the Russian Federation at the clinical site Publicly Funded, Krasnoyarsk, Krasnoyarsk Krai
  - State Funded Healthcare Institution of Moscow of City Health Department "V.M. Buyanov Municipal Clinical Hospital", Moscow, Moscow Oblast
  - Federal State Institution "V.I. Kulakov Research Center for Obstetrics, Gynecology, and Perinatology" of the Ministry of Healthcare and Social Development of the Russian Federation., Moscow, Moscow Oblast
  - State Educational Government-Financed Institution of Higher Professional Education "Kazan State Medical University" of the Ministry of Health of the Russian at the clinical site of Kazan Maternity Hospital No. 3 named after V.S. Gruzdev, Kazan', Tatarstan Republic
  - State Funded Health Care Institution "Bryansk Municipal Hospital No 1, Bryansk, The Bryansk Region
  - Federal State Educational Government-Financed Institution of Higher Education "Kemerovo State Medical University" of the Ministry of Healthcare of the Russian Federation at the clinical site of Kemerovo Oblast Publicly Funded Healthcare Institution "L.A., Kemerovo, The Kemerovo Region
  - Federal State Funded Healthcare Institution "L.G. Sokolov Federal Biomedical Agency Clinical Hospital No 122"., Saint Petersburg, The Leningrad Region
  - Federal State Funded Scientific Institution "Research Institute of Obstetrics, Gynecology and Reproductology named after D.O. Ott" of the Ministry of Healthcare of the Russian Federation, Saint Petersburg, The Leningrad Region
  - Moscow Oblast State Funded Healthcare Institution "Moscow Oblast Research Institute of Obstetrics and Gynecology", Moscow, The Moscow Region
  - State Funded Healthcare Institution of Moscow of City Health Department "Moscow Municipal Clinical Hospital No 31", Moscow, The Moscow Region
  - State Educational Government-Financed Institution of Higher Professional Education "Rostov State Medical University" of the Ministry of Healthcare of the Russian Federation at the clinical site of Obstetrics and Pediatrics Research Institute, Rostov-on-Don, The Rostov Region
  - Federal State Educational Government-Financed Institution of Higher Education "I.P. Pavlov Ryazan State Medical University" of the Ministry of Healthcare of the Russian Federation at the clinical site of State Funded Healthcare Institution "Municipal Clin, Ryazan, The Ryazan Region
  - Federal State Funded Healthcare Institution "Ural Research Institute of Maternal and Infant Care" of the Ministry of Healthcare of the Russian Federation, Yekaterinburg, The Sverdlovsk Region

REFERENCES:
- [Background] Miller JH, Weinberg RK, Canino NL, Klein NA, Soules MR. The pattern of infertility diagnoses in women of advanced reproductive age. Am J Obstet Gynecol. 1999 Oct;181(4):952-7. doi: 10.1016/s0002-9378(99)70331-5. PMID 10521760
- [Background] Dun EC, Nezhat CH. Tubal factor infertility: diagnosis and management in the era of assisted reproductive technology. Obstet Gynecol Clin North Am. 2012 Dec;39(4):551-66. doi: 10.1016/j.ogc.2012.09.006. PMID 23182560
- [Background] Westrom L. Effect of acute pelvic inflammatory disease on fertility. Am J Obstet Gynecol. 1975 Mar 1;121(5):707-13. doi: 10.1016/0002-9378(75)90477-9. PMID 123123
- [Background] Westrom LV. Sexually transmitted diseases and infertility. Sex Transm Dis. 1994 Mar-Apr;21(2 Suppl):S32-7. PMID 8042113
- [Background] Patil M. Assessing tubal damage. J Hum Reprod Sci. 2009 Jan;2(1):2-11. doi: 10.4103/0974-1208.51335. PMID 19562067
- [Background] Sutherland AM. The changing pattern of tuberculosis of the female genital tract. A thirty year survey. Arch Gynecol. 1983;234(2):95-101. doi: 10.1007/BF00207681. PMID 6667046
- [Background] Mueller BA, Daling JR, Moore DE, Weiss NS, Spadoni LR, Stadel BV, Soules MR. Appendectomy and the risk of tubal infertility. N Engl J Med. 1986 Dec 11;315(24):1506-8. doi: 10.1056/NEJM198612113152402. PMID 3785307
- [Background] Schwartz L, Diamond M. Formation, Reduction, and Treatment of Adhesive Disease. Seminars in Reproductive Medicine. 1991; 9(02): p. 89-99.
- [Background] Vaid K, Mehra S, Verma M, Jain S, Sharma A, Bhaskaran S. Pan endoscopic approach "hysterolaparoscopy" as an initial procedure in selected infertile women. J Clin Diagn Res. 2014 Feb;8(2):95-8. doi: 10.7860/JCDR/2014/7271.4018. Epub 2014 Feb 3. PMID 24701493
- [Background] Neerja, Jain K. Role of laporoscopy-hysteroscopy in cases of infertility with pregnancy outcome. J Indian Med Assoc. 2014 Feb;112(2):85-6, 88. PMID 25935960
- [Background] Diamond MP, Daniell JF, Feste J, Surrey MW, McLaughlin DS, Friedman S, Vaughn WK, Martin DC. Adhesion reformation and de novo adhesion formation after reproductive pelvic surgery. Fertil Steril. 1987 May;47(5):864-6. doi: 10.1016/s0015-0282(16)59181-x. PMID 2952528
- [Background] DeCherney AH, Mezer HC. The nature of posttuboplasty pelvic adhesions as determined by early and late laparoscopy. Fertil Steril. 1984 Apr;41(4):643-6. doi: 10.1016/s0015-0282(16)47793-9. PMID 6231195
- [Background] Al-Jabri S, Tulandi T. Management and prevention of pelvic adhesions. Semin Reprod Med. 2011 Mar;29(2):130-7. doi: 10.1055/s-0031-1272475. Epub 2011 Mar 24. PMID 21437827
- [Background] Brochhausen C, Schmitt VH, Planck CN, Rajab TK, Hollemann D, Tapprich C, Kramer B, Wallwiener C, Hierlemann H, Zehbe R, Planck H, Kirkpatrick CJ. Current strategies and future perspectives for intraperitoneal adhesion prevention. J Gastrointest Surg. 2012 Jun;16(6):1256-74. doi: 10.1007/s11605-011-1819-9. PMID 22297658
- [Background] Coulthard LR, White DE, Jones DL, McDermott MF, Burchill SA. p38(MAPK): stress responses from molecular mechanisms to therapeutics. Trends Mol Med. 2009 Aug;15(8):369-79. doi: 10.1016/j.molmed.2009.06.005. Epub 2009 Aug 6. PMID 19665431
- [Background] Ward BC, Kavalukas S, Brugnano J, Barbul A, Panitch A. Peptide inhibitors of MK2 show promise for inhibition of abdominal adhesions. J Surg Res. 2011 Jul;169(1):e27-36. doi: 10.1016/j.jss.2011.01.043. Epub 2011 Feb 23. PMID 21492875
- [Background] Katada J, Saito H, Ohashi A. Significance of cyclooxygenase-2 induced via p38 mitogen-activated protein kinase in mechanical stimulus-induced peritoneal adhesion in mice. J Pharmacol Exp Ther. 2005 Apr;313(1):286-92. doi: 10.1124/jpet.104.078717. Epub 2004 Dec 2. PMID 15576468
- [Background] U.S. Food and Drug Administration. U.S. Food and Drug Administration. [Online]. Northborough; 2006 [cited 2015 Dec 22. Available from: http://www.fda.gov/ohrms/dockets/ac/06/briefing/2006-4217b1_01_Executive%20Summary.pdf.
- [Background] Ghonge NP, Ghonge SD. Computed tomography and magnetic resonance imaging in the evaluation of pelvic peritoneal adhesions: What radiologists need to know? Indian J Radiol Imaging. 2014 Apr;24(2):149-55. doi: 10.4103/0971-3026.134400. PMID 25024524
- [Background] diZerega GS. The peritoneum and its response to surgical injury. Prog Clin Biol Res. 1990;358:1-11. No abstract available. PMID 2217485
- [Background] diZerega GS, Campeau JD. Peritoneal repair and post-surgical adhesion formation. Hum Reprod Update. 2001 Nov-Dec;7(6):547-55. doi: 10.1093/humupd/7.6.547. PMID 11727863
- [Background] Lali FV, Hunt AE, Turner SJ, Foxwell BM. The pyridinyl imidazole inhibitor SB203580 blocks phosphoinositide-dependent protein kinase activity, protein kinase B phosphorylation, and retinoblastoma hyperphosphorylation in interleukin-2-stimulated T cells independently of p38 mitogen-activated protein kinase. J Biol Chem. 2000 Mar 10;275(10):7395-402. doi: 10.1074/jbc.275.10.7395. PMID 10702313
- [Background] Kumar B, Koul S, Petersen J, Khandrika L, Hwa JS, Meacham RB, Wilson S, Koul HK. p38 mitogen-activated protein kinase-driven MAPKAPK2 regulates invasion of bladder cancer by modulation of MMP-2 and MMP-9 activity. Cancer Res. 2010 Jan 15;70(2):832-41. doi: 10.1158/0008-5472.CAN-09-2918. Epub 2010 Jan 12. PMID 20068172
- [Background] Louizos AA, Hadzilia SJ, Leandros E, Kouroukli IK, Georgiou LG, Bramis JP. Postoperative pain relief after laparoscopic cholecystectomy: a placebo-controlled double-blind randomized trial of preincisional infiltration and intraperitoneal instillation of levobupivacaine 0.25%. Surg Endosc. 2005 Nov;19(11):1503-6. doi: 10.1007/s00464-005-3002-4. Epub 2005 Oct 3. PMID 16328673
- [Background] Innes A, Burden RP, Finch RG, Morgan AG. Treatment of resistant peritonitis in continuous ambulatory peritoneal dialysis with intraperitoneal urokinase: a double-blind clinical trial. Nephrol Dial Transplant. 1994;9(7):797-9. PMID 7970121
- [Background] Szem JW, Hydo L, Barie PS. A double-blinded evaluation of intraperitoneal bupivacaine vs saline for the reduction of postoperative pain and nausea after laparoscopic cholecystectomy. Surg Endosc. 1996 Jan;10(1):44-8. doi: 10.1007/s004649910011. PMID 8711605
- [Background] Labaille T, Mazoit JX, Paqueron X, Franco D, Benhamou D. The clinical efficacy and pharmacokinetics of intraperitoneal ropivacaine for laparoscopic cholecystectomy. Anesth Analg. 2002 Jan;94(1):100-5, table of contents. doi: 10.1097/00000539-200201000-00019. PMID 11772809
- [Background] Ahmad G, Mackie FL, Iles DA, O'Flynn H, Dias S, Metwally M, Watson A. Fluid and pharmacological agents for adhesion prevention after gynaecological surgery. Cochrane Database Syst Rev. 2014 Jul 9;(7):CD001298. doi: 10.1002/14651858.CD001298.pub4. PMID 25005450
- [Background] U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), Center for Biologics Evaluation and Research (CBER). Non-Inferiority Clinical Trials.; 2010 [cited 2015 Dec. Available from: http://www.fda.gov/downloads/Drugs/./Guidances/UCM202140.pdf.
- [Background] Chow S, Shao J, Wang H. Sample Size Calculations in Clinical Research. 2nd ed.: Chapman&Hall / CRC Biostatistics Series; 2008.
- [Background] Guerriero S, Ajossa S, Lai MP, Mais V, Paoletti AM, Melis GB. Transvaginal ultrasonography in the diagnosis of pelvic adhesions. Hum Reprod. 1997 Dec;12(12):2649-53. doi: 10.1093/humrep/12.12.2649. PMID 9455829
- [Background] Guerriero S, Ajossa S, Garau N, Alcazar JL, Mais V, Melis GB. Diagnosis of pelvic adhesions in patients with endometrioma: the role of transvaginal ultrasonography. Fertil Steril. 2010 Jul;94(2):742-6. doi: 10.1016/j.fertnstert.2009.03.035. Epub 2009 Apr 14. PMID 19368917
- [Background] Julious SA. Sample Sizes for Clinical Trials: CRC Press/Taylor & Francis; 2010.
- [Background] Gnoth C, Godehardt E, Frank-Herrmann P, Friol K, Tigges J, Freundl G. Definition and prevalence of subfertility and infertility. Hum Reprod. 2005 May;20(5):1144-7. doi: 10.1093/humrep/deh870. Epub 2005 Mar 31. PMID 15802321
- [Background] Gnoth C, Godehardt D, Godehardt E, Frank-Herrmann P, Freundl G. Time to pregnancy: results of the German prospective study and impact on the management of infertility. Hum Reprod. 2003 Sep;18(9):1959-66. doi: 10.1093/humrep/deg366. PMID 12923157

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 114 is the number of enrolled and screened participants according to the protocol, but during the screening process some people were withdrawn from the study before randomization because some of them did not meet the inclusion criteria and some withdrew the informed consent form themselves. So, the number of randomized participants is 104.
Period: Overall Study
Arm/Group | Placebo, 1.5 mL/kg | Placebo, 2.4 mL/kg | Seroguard, 1.5 mL/kg | Seroguard, 2.4 mL/kg
Started | 26 | 26 | 26 | 26
Completed | 25 | 25 | 25 | 26
Not Completed | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, 1.5 mL/kg | Placebo, 2.4 mL/kg | Seroguard, 1.5 mL/kg | Seroguard, 2.4 mL/kg | Total
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 26 | 26 | 26 | 104
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (6.2) | 31.6 (5.3) | 31.6 (5.4) | 31.6 (5.4) | 31.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 26 | 26 | 104
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian race | 26 | 26 | 26 | 26 | 104
Region of Enrollment [Number; unit: participants]
  Russia | 26 | 26 | 26 | 26 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction of Adhesions Number by 3 or More
Description: The number of adhesions according to the first MRI data was compared to the number according to the data of second MRI
Time Frame: 30±4 days after surgical intervention
Population: 7 patients had no results of repeated Pelvic MRI examination that is why the number of Participants is different
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo, 1.5 mL/kg | Placebo, 2.4 mL/kg | Seroguard, 1.5 mL/kg | Seroguard, 2.4 mL/kg
Number analyzed (Participants) | 24 | 25 | 23 | 25
Participants | 1 | 1 | 10 | 10

2. Secondary Outcome: Change in Thickness of Pelvic Adhesions
Description: The change from baseline was defined. It was evaluated by comparing baseline MRI data and repeated MRI data. Results were estimated according to scale from 0 to 3 where 0 - no adhesions, 1 - thin (filmy or filiform), 2 - marked, 3 - marked with an impaired passage through organs involved.
Time Frame: 30±4 days after surgery
Population: 7 patients had no results of repeated Pelvic MRI examination that is why the number of Participants is different
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Placebo, 1.5 mL/kg | Placebo, 2.4 mL/kg | Seroguard, 1.5 mL/kg | Seroguard, 2.4 mL/kg
Number analyzed (Participants) | 24 | 25 | 23 | 25
score on a scale | 0 [0 to 2] | 0 [0 to 1] | 0 [0 to 2] | 0 [0 to 2]

3. Secondary Outcome: Number of Participants With Detection of Pelvic Organs Limited Mobility
Description: The frequency was estimated based on transvaginal ultrasound results
Time Frame: 30±4 days after surgery
Measure: Number; unit: participants
Arm/Group | Placebo, 1.5 mL/kg | Placebo, 2.4 mL/kg | Seroguard, 1.5 mL/kg | Seroguard, 2.4 mL/kg
Number analyzed (Participants) | 26 | 26 | 26 | 26
participants | 4 | 4 | 0 | 2

4. Secondary Outcome: Number of Participants With Detection of Hyperechoic Linear Lesions Post Surgery
Description: The frequency was estimated based on transvaginal ultrasound results
Time Frame: 30±4 days after surgery
Measure: Number; unit: participants
Arm/Group | Placebo, 1.5 mL/kg | Placebo, 2.4 mL/kg | Seroguard, 1.5 mL/kg | Seroguard, 2.4 mL/kg
Number analyzed (Participants) | 26 | 26 | 26 | 26
participants | 3 | 2 | 1 | 3

5. Secondary Outcome: Change in Number of Participants in Detecting Pelvic Organs Limited Mobility
Description: Absolute change of count of participants was measured with detecting pelvic organs limited mobility from the baseline
Time Frame: 30±4 days after surgery
Measure: Number; unit: participants
Arm/Group | Placebo, 1.5 mL/kg | Placebo, 2.4 mL/kg | Seroguard, 1.5 mL/kg | Seroguard, 2.4 mL/kg
Number analyzed (Participants) | 26 | 26 | 26 | 26
participants | -17 | -17 | -21 | -21

6. Secondary Outcome: Change Number of Participants in Detecting Hyperechoic Linear Lesions
Description: Frequency of detecting after repeated transvaginal ultrasound results was compared to baseline indications (4 or more)
Time Frame: 30±4 days after surgery
Measure: Number; unit: participants
Arm/Group | Placebo, 1.5 mL/kg | Placebo, 2.4 mL/kg | Seroguard, 1.5 mL/kg | Seroguard, 2.4 mL/kg
Number analyzed (Participants) | 26 | 26 | 26 | 26
participants | -17 | -16 | -19 | -18

7. Secondary Outcome: Number of Participants With Detection of no Ultrasound Signs of Pelvic Adhesive Disease Post Surgery
Description: No limited mobility of pelvic organs and no hyperechoic linear lesions should be shown
Time Frame: 30±4 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo, 1.5 mL/kg | Placebo, 2.4 mL/kg | Seroguard, 1.5 mL/kg | Seroguard, 2.4 mL/kg
Number analyzed (Participants) | 26 | 26 | 26 | 26
Participants | 19 | 19 | 23 | 20

ADVERSE EVENTS:
Time Frame: 30+-4 days
Arm/Group | Placebo, 1.5 mL/kg | Placebo, 2.4 mL/kg | Seroguard, 1.5 mL/kg | Seroguard, 2.4 mL/kg
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 3/25 | 2/25 | 1/25 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, 1.5 mL/kg (N=25) | Placebo, 2.4 mL/kg (N=25) | Seroguard, 1.5 mL/kg (N=25) | Seroguard, 2.4 mL/kg (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polymenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03660787/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT03660787/SAP_001.pdf